CLINICAL TRIAL: NCT03054532
Title: Phase II Study of Durvalumab in Combination With Lenalidomide in Relapsed/Refractory NK-T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDBCC-LYM-16-01
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: LYMPHOMA
MeSH Terms: conditions — Lymphoma | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Open-label phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Durvalumab and lenalidomide (Experimental): Open-label use of 2 drugs:
  * Durvalumab 1500 mg intravenously on day 1 of a 28-day cycle until progressive disease or intolerance.
  * Lenalidomide orally on days 1 through 21 of each 28-day cycle for 6 cycles.
  Interventions: Drug: Durvalumab; Drug: Lenali

INTERVENTIONS:
Drug: Durvalumab — Durvalumab intravenous 1500 mg
Drug: Lenali — Lenalidomide oral 20 mg/day

SUMMARY:
This is a multi-center, open-label, phase II study of durvalumab in combination with lenalidomide for treatment of relapsed/refractory NK/T-cell lymphoma (NKTCL). The study will employ a 2-stage Simon Optimal design with 80% power and type 1 error rate (significance level) of 5%. Stage 1 will involve 8 patients and will require at least 2 patients to achieve the primary end point of overall response in order to proceed onto to stage 2, which will have a target enrolment of 14 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven NK/T-cell lymphoma that has relapsed after at least one cycle of induction chemotherapy.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
3. Previously treated with at least one cycle of chemotherapy that includes L-asparaginase or gemcitabine.
4. Must be aged ≥ 21 years and able to sign informed consent form.
5. Adequate hematological function (unless abnormalities are related to lymphoma infiltration of the bone marrow or hemophagocytic syndrome related to NKL) within 30 days prior to signing informed consent, including:

   1. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
   2. Platelet count ≥ 50 x 109/L
   3. Hemoglobin ≥ 8 g/dL
6. Must be able to adhere to study visit schedules and other protocol requirements.
7. Females of childbearing potential must:

   1. Have 2 negative pregnancy tests as verified by a Study Investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the patient practices complete abstinence from heterosexual contact.
   2. Either commit to complete abstinence from heterosexual contact or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting study drug, during the study therapy (including dose interruptions), and for 28 days after discontinuation of study therapy.
8. Male patients must practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or female of childbearing potential while participating in the study, during dose interruptions and for 28 days after discontinuation of study therapy, even if he has undergone successful vasectomy.
9. All patients must:

   1. Have an understanding that the study drug could have a potential teratogenic risk.
   2. Agree to abstain from donating blood while taking study drug, during dose interruptions and for 28 days after discontinuation of study therapy.
   3. Agree not to share study medication with another person.
   4. Agree to be counseled about pregnancy precautions and risk of fetal exposure.
   5. Females must agree to abstain from breast feeding during the study participation and for 28 days after discontinuation of study therapy.
10. Male subjects should not donate sperm or semen while taking lenalidomide, during breaks (dose interruptions), and for at least 28 days after the last dose of lenalidomide.

Exclusion Criteria:

1. Concomitant use of any other investigational agent.
2. Known infection with human immunodeficiency virus (HIV).
3. Patient has known clinically active hepatitis B; carriers of hepatitis B are permitted but need to be on appropriate anti-viral therapy or have regular hepatitis B DNA virus monitored as advised by a Gastroenterologist.
4. Subject has a calculated or measured creatinine clearance of < 30 mL/minute.
5. Neuropathy > Grade 2.
6. Presence of CNS involvement by lymphoma.
7. Myocardial infarction within 6 months prior to enrolment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
8. Clinically significant active infection or uncontrolled intercurrent illness.
9. Pregnant or lactating females.
10. Coexistent second malignancy or history of prior malignancy within the preceding 3 years (excluding non-melanoma skin tumors or in situ carcinoma of the cervix).
11. Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by overall response rate measured at the time of best response. | 2 years
  Overall response rate (ORR) is defined as the proportion of patients with reduction in tumor burden of at least 50%.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS is defined as the time from enrolment to progression or death due to any cause. The distribution of PFS will be estimated using the method of Kaplan-Meier.
Overall survival (OS) | 2 years
  OS is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time-to-response (TTR) | 2 years
  Defined for all evaluable patients who have achieved an overall response as the date at which the patient's objective status is first noted to be a CR or PR.
Duration of response (DoR) | 2 years
  Defined for all evaluable patients who have achieved an overall response as the date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression is documented.

CONTACTS AND LOCATIONS:
Locations (4):
- Singapore (4):
  - National University Hospital Singapore, Singapore
  - Singapore General Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
  - Raffles Hospital Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No